CLINICAL TRIAL: NCT04076462
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Multi-center Trial to Assess Efficacy and Safety of Octreotide Subcutaneous Depot (CAM2029) in Patients With Acromegaly
Brief Title: A Trial to Assess Efficacy and Safety of Octreotide Subcutaneous Depot in Patients With Acromegaly
Acronym: ACROINNOVA 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Camurus AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HS-18-633; 2019-001191-11 (EudraCT Number)
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Acromegaly
Keywords: Acromegaly; octreotide; CAM2029; phase 3
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CAM2029 (octreotide subcutaneous depot) (Experimental): CAM2029 (octreotide subcutaneous depot) 20mg/1.0 mL for 20 mg dose, subcutaneous injection once monthly, six months treatment. If down-titration is required, 10mg/0.5 mL for 10 mg dose is available.
  Interventions: Drug: CAM2029 (octreotide subcutaneous depot)
- Matching placebo (Placebo Comparator): Placebo (subcutaneous depot) 1.0 mL, subcutaneous injection once monthly, six months treatment. If down-titration is required, 0.5 mL dose is available.
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: CAM2029 (octreotide subcutaneous depot) — Octreotide subcutaneous depot for monthly injections in acromegaly patients
  Other Names: CAM2029
  Arms: CAM2029 (octreotide subcutaneous depot)
Drug: Matching placebo — Matching placebo for CAM2029
  Other Names: placebo
  Arms: Matching placebo

SUMMARY:
The purpose of this trial is to assess the efficacy and safety of CAM2029 in patients with acromegaly. Patients will be randomized to either CAM2029 or placebo administered subcutaneously once monthly during 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, ≥18 years at screening
* Able to provide written informed consent to participate in the trial prior to any trial related procedures are performed
* Diagnosis of acromegaly by historical evidence of (persistent or recurrent) acromegaly
* Treatment with a stable dose of octreotide LAR or lanreotide ATG for at least 3 months as monotherapy prior to screening
* IGF-1 levels ≤1xULN at screening
* Adequate liver, pancreatic, renal and bone marrow functions
* Normal ECG

Exclusion Criteria:

* GH ≥2.5 μg/L at screening (cycle)
* Have received medical treatment for acromegaly with pasireotide (within 6 months prior to screening), pegvisomant (within 3 months prior to screening), dopamine agonists (within 3 months prior to screening) or other investigational agents (within 30 days or 5 half-lives prior to screening [whichever is longer]
* Patients who usually take octreotide LAR or lanreotide ATG less frequently than every 4 weeks (e.g. every 6 weeks or 8 weeks)
* Patients with compression of the optic chiasm causing any visual field defect for whom surgical intervention is indicated
* Patients who have undergone major surgery/surgical therapy for any cause within 1 month from screening
* Patients who have undergone pituitary surgery within 6 months prior to screening
* Patients who have received prior pituitary irradiation
* Patients with poorly controlled diabetes mellitus (hemoglobin A1c >8.0%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with mean IGF-1 levels ≤1xULN | Week 22 and 24

SECONDARY OUTCOMES:
Proportion of patients with mean IGF-1 levels ≤1xULN, including patients with dose reduction | Week 22 and 24
Proportion of patients with mean IGF-1 levels ≤1xULN at Week 22/Week 24 and mean GH levels <2.5 µg/L at Week 24 | Week 22 and 24
Proportion of patients with mean GH levels <2.5 µg/L | Week 24
Proportion of patients with mean GH levels <1.0 µg/L | Week 24
Incidence of treatment emergent adverse events | Week 0 to 24
Proportion of patients/partners declared competent by a healthcare professional to administer intervention | Week 0 to 20 and week 24
  During patients/partners first three attempts during the trial period of 24 weeks whenever these visits take place
Octreotide plasma concentrations over time | Week 0 to 24

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Freda, M.D, Principal Investigator — Columbia University
Locations (63):
- United States (12):
  - UCLA Department of Medicine Division of Endocrinology, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - Prufen Clinical Research LLC, Miami, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University in St. Louis, School of Medicine, St Louis, Missouri
  - Palm Research Center, Las Vegas, Nevada
  - Columbia University Medical Center, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Allegheny Endocrinology Associates, Pittsburgh, Pennsylvania
  - Research Institute of Dallas, Dallas, Texas
- Germany (6):
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Frankfurt, Medizinische Klinik 1, Schwerpunkt Endokrinologie, Diabetologie, Ernährungsmedizin, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - LMU Clinic of University of Munich, Medical Clinic and Polyclinic IV, Munich
  - Medicover Neuroendokrinologie, Munich
  - Medicover Oldenburg MVZ, Oldenburg
- Greece (3):
  - General Hospital of Athens "Laiko", Endocrinology University Clinic, Athens
  - Aretaeio University Hospital Endocrinology Department, Faculty of Diabetes and Metabolism, Athens
  - General Hospital of Thessaloniki "Ippokratio", Thessaloniki
- Hungary (2):
  - Military Healt Center, 2nd Department of Internal Medicine, Budapest
  - SZTE ÁOK I.sz. Belgyógyászati Klinika, Szeged
- Italy (5):
  - IRCCS Policlinico San Martino, Genova
  - Azienda Universitaria "Federico II", Napoli
  - Azienda Ospedaliera Padova, Department of Internal medicine, Padua
  - Policlinic Gemelli University Hospital IRCCS, Department of Endocrinology, Roma
  - AOUI Verona, Policlinic of GB Rossi, Verona
- Poland (4):
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Szpital Uniwersytecki w Krakowie, Krakow
  - Centrum Nowoczesnych Terapii "Dobry Lekarz", Krakow
  - Amicare Sp. z o.o. Sp. K., Lodz
  - Piekarskie Centrum Medyczne, Szpital Miejski, Piekary Śląskie
- Russia (7):
  - Interregional Clinical Diagnostic Center, Kazan'
  - "Atlas" Medical Center, Moscow
  - Sechenov Moscow First State Medical University, Moscow
  - Vladimirsky Moscow Regional Research Clinical Institute, Moscow
  - Novosibirsk State Regional Clinical Hospital, Novosibirsk
  - Interregional Clinical Diagnostic Center, Ryazan
  - Saratov Regional Clinic Hospital, Saratov
- Spain (9):
  - University Hospital Complex A Coruña, A Coruña
  - University Hospital of Alicante, Alicante
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid
  - Complejo Hospitalario Universitario Santiago de Compostela, Santiago de Compostela
  - University Hospital Virgen del Rocio, Seville
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Universitario de la Ribera, Valencia
- Turkey (Türkiye) (10):
  - Akdeniz University Faculty of Medicine Department of Endocrinology, Antalya
  - Aydın Adnan Menderes University Research and Application Hospital, Aydin
  - Pamukkale University Faculty of Medicine Department of Endocrinology, Denizli
  - Eskisehir Osmangazi University Medical Faculty, Eskişehir
  - Istanbul University Medical Faculty, Fatih
  - Kocaeli University Faculty of Medicine Department of Endocrinology and Metabolism, Kocaeli
  - Inonu University Medical Faculty Endocrinology Department, Malatya
  - Erciyes University Medical Faculty, Dept. of Endocrinology, Melikgazi
  - Karadeniz Technical University Farabi Hospital, Trabzon
  - Zonguldak Bulent Ecevit University Department of Internal Medicine, Division of Endocrinology and Metabolism Ibni Sina Campus, Zonguldak
- United Kingdom (5):
  - College of Medical and Dental Sciences, Birmingham
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - The Christie NHS Foundation Trust, Manchester
  - Salford Royal Foundation Trust, Salford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Glatard A, Friberg-Hietala S, Keutzer L, Hansson A, Johnsson M, Tiberg F. Population Pharmacokinetic Analysis of an Octreotide Depot (CAM2029) in the Treatment of Acromegaly. Clin Pharmacokinet. 2025 Jul;64(7):1079-1092. doi: 10.1007/s40262-025-01522-3. Epub 2025 May 26. PMID 40418492
- [Derived] Ferone D, Freda P, Katznelson L, Gatto F, Kadioglu P, Maffei P, Seufert J, Silverstein JM, Spencer-Segal JL, Isaeva E, Dreval A, Harrie M, Svedberg A, Tiberg F. Octreotide Subcutaneous Depot for Acromegaly: A Randomized, Double-blind, Placebo-controlled Phase 3 Trial, ACROINNOVA 1. J Clin Endocrinol Metab. 2025 May 19;110(6):1729-1739. doi: 10.1210/clinem/dgae707. PMID 39378125